CLINICAL TRIAL: NCT04941417
Title: Neoadjuvant Immunotherapy With Chemotherapy for the Treatment of Stage I-IIIB Non-Small Cell Lung Cancer (NSCLC): A Phase II Exploratory Study
Brief Title: Neoadjuvant Immunotherapy With Chemotherapy for Stage I-IIIB Non-Small Cell Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Junling Li, Professor, Peking Union Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2873
Record Dates: First submitted 2021-05-17; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant PD-(L)1 inhibitor with chemotherapy followed by PD-(L)1 inhibitor for up to 1 year (Experimental)
  Interventions: Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: PD-1 inhibitor — Two to three cycles of neoadjuvant chemotherapy in combination with PD-(L)1 inhibitor will be administered before surgery, followed by another one to two cycles of neoadjuvant chemotherapy in combination with PD-(L)1 inhibitor and PD-(L)1 inhibitor monotherapy for up to 1 year.

SUMMARY:
A phase II, single-arm, open-label study that assesses feasibility, safety and efficacy of combined neoadjuvant chemotherapy and immunotherapy with PD-(L)1 inhibitor in stage I-IIIB NSCLC adult patients followed by adjuvant PD-(L)1 inhibitor treatment for up to 1 year

DETAILED DESCRIPTION:
A phase II, single-arm, open-label study that assesses feasibility, safety and efficacy of combined neoadjuvant chemotherapy and immunotherapy with PD-1 inhibitor in stage I-IIIB NSCLC adult patients followed by adjuvant treatment for up to 1 year with PD-(L)1 inhibitor.

Two to three cycles of neoadjuvant chemotherapy in combination with PD-(L)1 inhibitor will be administered before surgery, followed by another one to two cycles of neoadjuvant chemotherapy in combination with PD-(L)1 inhibitor and PD-(L)1 inhibitor monotherapy for up to 1 year.

After completion of neoadjuvant therapy and before surgery, a tumor assessment will be done. Patients with stable disease or partial response may be considered for surgery.

The report imaging response and pathological response rate will be evaluated. Patients eligible for the trial are those with a histological diagnosis or cytologically proven operable and resectable non-small-cell lung cancer. The total number of patients to be included will be 60 from Chinese Academy of Medical Sciences (CAMS).

Accrual period of 2 years or until the inclusion of the last patient necessary to achieve the sample set in the protocol of 60 patients. After that all patients will be treated for up to 1 year with adjuvant immunotherapy and they will be followed during 3 years after adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

- 1.Histologically- or cytologically- documented NSCLC who present stage I (T≥4cm), IIA, IIB, IIIA, or IIIB disease, of either squamous or non-squamous histology.

2.Deemed surgically resectable by a thoracic surgeon 3.Age ≥ 18 years 4.Radiologically measurable disease, as defined by response evaluation criteria in solid tumours (RECIST) v1.1 5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 6.Notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines.

Exclusion Criteria:

* 1. Carrying activating mutations in the TK domain of EGFR or any variety of alterations in the ALK gene or other mutations predicting hyperprogression of immunotherapy.

  2. Active, known or suspected autoimmune disease. 3.Other active malignancy requiring concurrent intervention or with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast).

  4.Prior treatment with anti-PD-1, anti-CTLA-4 (cytotoxic T lymphocyte-associated antigen (CTLA-4), or anti-PD-L1 therapeutic antibody or pathway-targeting agents 5.History of allergy to study drug components excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
MPR (major pathologic response) | Up to 8 weeks
  Major pathologic response (MPR) is defined as > 90 percent decrease in viable tumor.

SECONDARY OUTCOMES:
DFS(disease-free survival) | at 3 years from the first dose of neoadjuvant treatment
  Time from first dose of neoadjuvant treatment to recurrence of tumor or death
OS(overall survival) | at 3 years from the first dose of neoadjuvant treatment
  Time when the patient is still alive
Toxicity profile | from the first dose of neoadjuvant treatment until 90 days after the last dose of adjuvant treatment
  Toxicities caused by the drug during the study，according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No